CLINICAL TRIAL: NCT05146167
Title: Reducing HIV/Sexually Transmitted Infection (STI) Risk Behaviors Among Juvenile Offenders on Probation: A Mobile Mindfulness-Based Intervention
Brief Title: Feasibility Testing a Meditation App for Youth in the Legal System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ashley D Kendall, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-0889; R00DA047890 (NIH)
Record Dates: First submitted 2021-11-08; First posted 2021-12-06 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-04

CONDITIONS: Behavioral Health
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be individually randomized at a 1:1 ratio to 1 of 2 smartphone app conditions: (1) Bodhi AIM (Action In Mindfulness), a 30-day meditation app, or (2) HIB (Health In Balance), a health promotion control app matched to Bodhi AIM for time and structure.
Who Masked: Outcomes Assessor
Masking Description: Both participants and outcome assessors will be blind to condition through completion of the baseline assessment. Condition will become apparent to both participants and assessors at the time of app download, but will not be revealed to assessors at either of the follow-up time points until after the quantitative measures are complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bodhi AIM (Experimental): Participants randomized to the intervention arm will receive the Bodhi AIM meditation app.
  Interventions: Behavioral: Bodhi AIM (intervention group)
- HIB (Active Comparator): Participants randomized to the active control arm will receive the HIB health promotion app.
  Interventions: Behavioral: HIB (control group)

INTERVENTIONS:
Behavioral: Bodhi AIM (intervention group) — Bodhi AIM (Action In Mindfulness) is a smartphone-based app that teaches users to establish a daily meditation practice via a 30-day "path," with each day consisting of a brief audio- or video-guided file. In addition to the 30 daily path files, users have access to a menu of "to go" audio-guided meditation practices that they may access any time to prepare for particular situations (e.g., attending a party).
  Arms: Bodhi AIM
Behavioral: HIB (control group) — HIB (Health In Balance) is a smartphone-based app that is matched to Bodhi AIM for time and structure, but includes health promotion content (e.g., educational information on substance use) in place of the meditation content featured in Bodhi AIM. Like Bodhi AIM, HIB includes a 30-day "path" of audio and video files, along with a menu of "to go" audio files that users may access any time to review key intervention concepts.
  Arms: HIB

SUMMARY:
This feasibility clinical trial aims to assess the feasibility of implementing a 1-month app-based meditation program with youth in the juvenile legal system. The primary questions it is designed to answer are:

1. Will youth adequately adhere to the 1-month meditation app?
2. Is it feasible to collect data remotely from youth on their self-reported cannabis use, sexual health, and mental health at baseline, 1, and 6 months?

DETAILED DESCRIPTION:
The investigators aim enroll 100 youth in Cook County, IL 13-18 years old who report regular access to an Apple or Android smartphone. Following completion of a baseline questionnaire, participants will be individually randomized at a 1:1 ratio to 1 of 2 smartphone app conditions: (1) Bodhi AIM (Action In Mindfulness), a 30-day meditation app or (2) HIB (Health In Balance), a health promotion control app matched to Bodhi AIM for time and structure. Follow-up assessments will occur at 1 and 6 months. All study activities will be remote.

ELIGIBILITY:
Inclusion Criteria:

* 13-18 years old
* In probation programming (i.e., in legal programming but not detained) in Cook County, IL
* Have access to an Apple/Android smartphone
* Understand and provide assent/consent
* Have legal guardian permission (if under 18 years old)
* English-speaking, due to norming of instruments

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 107 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
App adherence | 1 month
  Days of objective app usage
Percentage of participants who complete the cannabis use measure at each time point | Baseline, 1 month, 6 months
  Cannabis use is measured with the Cannabis Use Disorders Identification Test-Revised
Percentage of participants who complete the sexual health measure at each time point | Baseline, 1 month, 6 months
  Sexual health is measured with a modified version of the AIDS Risk Behavior Assessment
Percentage of participants who complete the mental health symptoms measure at each time point | Baseline, 1 month, 6 months
  Mental health symptoms are measured with the Youth Self Report

SECONDARY OUTCOMES:
Percentage of participants who complete other substance use measures at each time point | Baseline, 1 month, 6 months
  The other substance use measures include the Young Adult Alcohol Problem Scale, the Alcohol Trouble Scale, the Hangover Symptoms Scale, and a modified Substance Use Self-Efficacy Scale
Percentage of participants who complete other mental health measures at each time point | Baseline, 1 month, 6 months
  The other mental health measures include the Reactive-Proactive Aggression Questionnaire, the Short-Form Buss-Perry Aggression Questionnaire, the Negative Mood Regulation Scale, the Connor-Davidson Resilience Scale-10, and the Five Facets of Mindfulness Questionnaire-15

OTHER OUTCOMES:
Percentage of participants who complete other outcome measures at each time point | Baseline, 1 month, 6 months
  The other outcome measures include self-reported legal system involvement (e.g., frequencies of arrests and detainments), the UCLA PTSD Rating Index, and the Digital Working Alliance Inventory (measured at 1 month and 6 months only)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley D Kendall, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be made available upon reasonable request.